CLINICAL TRIAL: NCT01117168
Title: Protocol for the Enrollment on the Official COG Registry, The Childhood Cancer Research Network (CCRN)
Brief Title: Enrollment on the Childhood Cancer Research Network (CCRN) of the Children's Oncology Group
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACCRN07; 10-C-0111; 100111 (Other: National Cancer Institute (NCI)); NCT00799253 (obsolete NCT alias)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Cancer; Leukemia; Sarcoma; Brain Tumors
Keywords: Children's Oncology Group; Pediatric Oncology; Pediatric Cancer; Registration; Leukemia; Brain Tumor; Sarcoma
MeSH Terms: conditions — Neoplasms; Leukemia; Sarcoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The Children's Oncology Group has established a research network, the Childhood Cancer Research Network (CCRN), to collect information about children with cancer and other conditions that are benign but involve abnormal cell growth in order to help doctors and scientists better understand childhood cancer. The CCRN's goal is to collect clinical information about every child diagnosed with cancer and similar conditions in the United States and Canada, to allow researchers to study patterns, characteristics, and causes of childhood cancer. The information can also help researchers study the causes of childhood cancer. To expand the CCRN, parents of children who have been diagnosed with cancer will be asked to provide information about themselves and their child for research purposes.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To obtain informed consent from parents of infants, children, adolescents, and young adults newly diagnosed with cancer (and their child when appropriate) to enter their names and certain information concerning their child into the Childhood Cancer Research Network and/or for permission to be contacted in the future to consider participating in future studies.

II. For children under the age of majority at the time of parental consent: Once the child reaches the age of majority, to obtain informed consent from that child to allow her/his name and other identifying information to continue to be available to the Childhood Cancer Research Network and/or to be possibly contacted in the future to consider participating in other studies.

OUTLINE:

Institutional membership in the Children's Oncology Group (COG) requires registration of all pediatric cancer patients seen at their site. This registration process includes all patients. In order to maximize the resource that a network would provide, it is necessary to have identifying information on a large proportion of the cases included within the network. Moreover, the resource would be further enhanced if informed consent from parents/patients was obtained to allow future contact regarding possible participation in non-therapeutic and prevention research.

ELIGIBILITY:
* All patients, diagnosed with a primary malignancy since the date the initial IRB approval was received for this study with any of the following diagnoses are eligible:
* All cancer cases with an ICD-O histologic behavior code of two "2" (carcinoma in situ) or three "3" (malignant).
* All lesions of the central nervous system regardless of behavior, i.e., benign, borderline or malignant.
* The benign/borderline conditions which will be reportable by agreement shall include:
* Mesoblastic nephroma.
* All teratomas, regardless of locations.
* Myeloproliferative disease
* Langerhans Cell histiocytosis
* Patients with a secondary malignancy may be eligible provided they also meet the criteria in the above. These patients need to be enrolled using their primary diagnosis.
* Participants 0 through 21 years of age are eligible; irrespective of eligibility for other COG studies.
* Participant must be resident of the United States, Canada or Mexico.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and adolescent patients diagnosed with cancer
Enrollment: 57816 (Actual)
Dates: Start 2010-04-30; Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To collect information on children with cancer | After initial diagnosis

SECONDARY OUTCOMES:
To obtain consent to contact in the future for participation in future clinical trials | At enrollment and at age of majority

CONTACTS AND LOCATIONS:
Overall Officials: Logan Spector, Study Chair; Susan Stork, CCRP, Study Chair
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Background] Ross JA, Severson RK, Pollock BH, Robison LL. Childhood cancer in the United States. A geographical analysis of cases from the Pediatric Cooperative Clinical Trials groups. Cancer. 1996 Jan 1;77(1):201-7. doi: 10.1002/(SICI)1097-0142(19960101)77:13.0.CO;2-7. PMID 8630931